CLINICAL TRIAL: NCT01102894
Title: Measurement of Whole Gut Transit Time After a Dietary Fiber Treatment Using a Wireless Motility Capsule
Brief Title: Pilot Study Using a Wireless Motility Capsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 0903M60781
Record Dates: First submitted 2010-03-24; First posted 2010-04-13 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low fiber and High Fiber (Experimental): Subjects consume a low fiber cereal and swallow the SmartPill device that measures gastrointestinal transit time Subjects consume a high fiber cereal along with swallowing the SmartPill device that measures gastrointestinal transit time
  Interventions: Device: SmartPill

INTERVENTIONS:
Device: SmartPill — SmartPill

SUMMARY:
Research suggests dietary fiber may decrease transit time through the gastrointestinal tract. Research studies traditionally use radio-opaque markers to determine gastric emptying, colonic transit, and whole gut transit time. The SmartPill is a single use pill that can be used to determine gastric emptying, colonic transit, and whole gut transit time without requiring X-rays or fecal collections. Previous studies have found radio-opaque markers and the SmartPill detect the similar transit times.

The purpose of this pilot study is to determine if the SmartPill can detect a change in transit time using a significant dose of dietary fiber.

DETAILED DESCRIPTION:
The ability of a device to track gastrointestinal transit time, including gastric emptying time, was measured in healthy people consuming low and high fiber diets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18 - 65
* Non-smoking
* Not taking medication
* Non-dieting
* BMI 18-30
* English literacy
* Ability to swallow the SmartPill

Exclusion Criteria:

* Do not regularly consume breakfast
* Food allergies to ingredients fond in study products
* Dislike of hot cereal
* BMI <18 or >30
* Are not weight stable
* Diagnosed with diabetes, cardiovascular, renal, or hepatic disease
* Cancer in previous 5 years (except basal cell carinoma of the skin)
* Any gastrointestinal disease or condition
* Any gastrointestinal surgeries that alter motility
* Recent antibiotic usage (< 6 months)
* recent or concurrent participation in an intervention research study
* History of drug or alcohol abuse in prior 6 months
* Use of laxatives, anti-diarrheal, antacids, or medications which alter motility
* Vegetarians
* People who eat more than approximately 15 grams of fiber per day
* Currently consume fiber supplements
* Women who are pregnant or lactating
* Women with irregular menstrual cycles

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - McNeal Hall, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Timm D, Willis H, Thomas W, Sanders L, Boileau T, Slavin J. The use of a wireless motility device (SmartPill(R)) for the measurement of gastrointestinal transit time after a dietary fibre intervention. Br J Nutr. 2011 May;105(9):1337-42. doi: 10.1017/S0007114510004988. Epub 2010 Dec 8. PMID 21138605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the University of Minnesota via fliers on the St. Paul campus
Pre-assignment Details: Exclusion criteria included contraindicated conditions for the SmartPill: dysphasia, gastric bezoars, strictures, fistulas, bowel obstructions, diverticulitis, previous gastrointestinal surgery, implanted electro-mechanical medical devices, and medications shown to influence gastrointestinal transit time.
Groups:
- High Fiber and Low Fiber: Subjects consume a low and high fiber cereal along with swallowing the SmartPill device that measures gastrointestinal transit time
  SmartPill : SmartPill
Period: Overall Study
Arm/Group | High Fiber and Low Fiber
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Fiber and High Fiber: Subjects consume a high fiber cereal along with swallowing the SmartPill device that measures gastrointestinal transit time Subjects also consumed low fiber
  SmartPill : SmartPill
Arm/Group | Low Fiber and High Fiber
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Whole Gut Transit Time
Description: The time required for the SmartPill to travel through the entire gastrointestinal tract and be present in the feces.
Time Frame: 5 days
Population: All participants had their transit time assessed.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- High Fiber: Subjects consume a high fiber cereal along with swallowing the SmartPill device that measures gastrointestinal transit time
  SmartPill : SmartPill
- Low Fiber: Subjects consume a low fiber cereal and swallow the SmartPill device that measures gastrointestinal transit time
  SmartPill : SmartPill
Arm/Group | High Fiber | Low Fiber
Number analyzed (Participants) | 10 | 10
hours | 22.5 (14.6) | 31.4 (5.8)

2. Secondary Outcome: Gastrointestinal Tolerance
Description: Subjects scored their gastrointestinal tolerance based on 7 questions on a 0-10 scale on day 4 of each treatment period and the sum score was reported. 0 being the best and 10 being the worst. Each question has a value of 1-10 for a total of 70 points as value.
Time Frame: Day 4
Population: Each participant completed a gastrointestinal tolerance questionnaire during each treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Fiber | Low Fiber
Number analyzed (Participants) | 10 | 10
units on a scale | 9.5 (1.7) | 6.8 (1.7)

3. Secondary Outcome: Food Intake Diary
Description: Total dietary fiber consumed.
Time Frame: Day 1
Population: Day 1 of each treatment subjects completed a 24 hour food record to determine baseline dietary fiber intake
Measure: Mean (Standard Deviation); unit: g
Arm/Group | High Fiber | Low Fiber
Number analyzed (Participants) | 10 | 10
g | 14 (7.5) | 15 (7)

ADVERSE EVENTS:
Time Frame: Study length
Description: No Adverse events were recorded during the study
Arm/Group | High Fiber | Low Fiber
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The study interventions were not randomized, which doesn't allow for period effect calculations. The SmartPill can reside in the stomach for longer than a few hours, which can skew results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No